CLINICAL TRIAL: NCT04583371
Title: Effect of the Use of Pulmonary Hyperinflation With Mechanical Ventilator Plus Aspiration Versus Isolated Tracheal Aspiration in Bronchial Hygiene in Patients With Heart Disease
Brief Title: The Use of Pulmonary Hyperinflation With the Mechanical Ventilator in Cardiac Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Bruna Eibel, PhD, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HPMVSASP
Record Dates: First submitted 2020-09-29; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Heart Diseases
Keywords: PHYSIOTHERAPY; Mechanical Ventilation
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: This is a randomized crossover clinical trial in which the individuals selected for the study will be randomized to receive isolated tracheal aspiration (Control Group) and pulmonary hyperinflation through the mechanical ventilator associated with tracheal aspiration (Intervention Group). Randomization will be performed through the randomization.com website by a 1: 1 crossed block, allocating the patient to one of the groups and, after 24 hours, another technique will be performed. In addition, a control aspiration will be performed 2 hours before both techniques.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP CONTROL (No Intervention): For basal aspiration, the patient will be placed in the supine position with the head elevated at 30º, will be submitted to a single aspiration with a size 12 probe (Mark Med), with a vacuum adjusted to -40cmH2O of pressure, with basic asepsis care being maintained for performing the technique.
  In the control group, patients will be ventilated for 1 minute with 100% inspired oxygen (FiO2), followed by three aspirations for 15 seconds and with an interval of 30 seconds.
- INTERVENTION GROUP (Active Comparator): For basal aspiration, the patient will be placed in the supine position with the head elevated at 30º, will be submitted to a single aspiration with a size 12 probe (Mark Med), with a vacuum adjusted to -40cmH2O of pressure, with basic asepsis care being maintained for performing the technique.
  In the participants of the intervention group, the calculation of the ideal tidal volume of each patient will be performed, after which they will be positioned in the supine position, the headboard elevated to 30º in assisted pressure-controlled ventilatory mode, increasing 10 cmH2O in inspiratory pressure and in assisted ventilation mode. -controlled by volume, we will increase 50% of the tidal volume for a period of 10 minutes, with Ppeak not exceeding 40 cmH2O and drive pressure not exceeding 15 cmH2O in both ventilation modes, and then a new aspiration in the same way as the control group.
  Interventions: Other: MECHANICAL PULMONARY HYPERINFLUATION

INTERVENTIONS:
Other: MECHANICAL PULMONARY HYPERINFLUATION — For basal aspiration, the patient will be placed in the supine position with the head elevated at 30º, will be submitted to a single aspiration with a size 12 probe (Mark Med), with a vacuum adjusted to -40cmH2O of pressure, with basic asepsis care being maintained for performing the technique. In the participants of the intervention group, the calculation of the ideal tidal volume of each patient will be performed, after which they will be positioned in the same way as baseline aspiration, in assisted-controlled pressure ventilation, increasing 10 cmH2O in inspiratory pressure and, in ventilatory mode. -controlled by volume, we will increase 50% of the tidal volume for a period of 10 minutes, observing the peak that cannot exceed 40 cmH2O in both ventilation modes, and then three aspirations will be performed for 15 seconds and with an interval of 30 seconds.
  Arms: INTERVENTION GROUP

SUMMARY:
Mechanical ventilation (MV) is used to reduce work and reverse or prevent fatigue of the respiratory muscles, decrease oxygen consumption and maintain gas exchange. In addition to the benefits given to patients undergoing MV, there is a high risk of accumulating bronchial secretions, related to pathology and / or therapeutic intervention. Pulmonary hyperinflation is widespread in patients in intensive care centers (ICUs) as a bronchial hygiene therapy, being used in 40% of 64 Australian ICUs as demonstrated by Dennis et al., Through contact with physical therapists. Mechanical hyperinflation associated with tracheal aspiration is able to increase the amount of secretion aspirated when compared to isolated aspiration in patients undergoing mechanical ventilation. To assess whether the pulmonary hyperinflation maneuver with the mechanical ventilator, compared to isolated tracheal aspiration, increases the removal of secretions. To evaluate whether the use of the pulmonary hyperinflation maneuver in the mechanical ventilator is hemodynamically stable through the collection in two moments of the variables of heart rate (HR), mean arterial pressure (MAP), peripheral saturation (SpO2), respiratory rate (RF) that will be analyzed from the postoperative unit's multiparametric monitor.

Evaluate the change in respiratory mechanics through collection in two moments after the mechanical hyperinflation technique through dynamic compliance (Cdyn), tidal air volume (VAC), peak pressure (Ppico). The population will consist of patients from the Post-Operative Unit (UPO), from the Institute of Cardiology, of both sexes, over 18 years old, mechanically ventilated and the sample consisting of 50 individuals. These will be submitted to the use of the pulmonary hyperinflation maneuver in the mechanical ventilator. Randomized crossover clinical trial.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) is used to reduce work and reverse or prevent fatigue of the respiratory muscles, decrease oxygen consumption and maintain gas exchange. In addition to the benefits given to patients undergoing MV, there is a high risk of accumulating bronchial secretions, related to pathology and / or therapeutic intervention. Pulmonary hyperinflation is widespread in patients in intensive care centers (ICUs) as a bronchial hygiene therapy, being used in 40% of 64 Australian ICUs as demonstrated by Dennis et al., Through contact with physical therapists. Mechanical hyperinflation associated with tracheal aspiration is able to increase the amount of secretion aspirated when compared to isolated aspiration in patients undergoing mechanical ventilation.

To evaluate whether the use of the pulmonary hyperinflation maneuver in the mechanical ventilator is hemodynamically stable through the collection in two moments of the heart rate (HR), mean arterial pressure (MAP), peripheral saturation (SpO2), respiratory rate (RF) variables that will be analyzed from the postoperative unit's multiparametric monitor.

Evaluate the change in respiratory mechanics through collection in two moments after the mechanical hyperinflation technique through dynamic compliance (Cdyn), tidal air volume (VAC), peak pressure (Ppico). The population will consist of patients from the Post-Operative Unit (UPO), unit intensive care (UCI) and emergency room, from the Institute of Cardiology, of both sexes, over 18 years old, mechanically ventilated more than 48 hours and the sample consisting of 50 individuals. These will be submitted to the use of the pulmonary hyperinflation maneuver in the mechanical ventilator.

This is a randomized crossover clinical trial in which the individuals selected for the study will be randomized to receive isolated tracheal aspiration (Control Group) and pulmonary hyperinflation through the mechanical ventilator associated with tracheal aspiration (Intervention Group). Randomization will be performed through the randomization.com website by a 1: 1 crossed block, allocating the patient to one of the groups and, after 24 hours, another technique will be performed. In addition, a control aspiration will be performed 2 hours before both techniques.

For basal aspiration, the patient will be placed in the supine position with the head elevated at 30º, will be submitted to a single aspiration with a size 12 probe (Mark Med), with a vacuum adjusted to -40cmH2O of pressure, with basic asepsis care being maintained for performing the technique35.

In the control group, patients will be ventilated for 1 minute with 100% inspired oxygen (FiO2), followed by three aspirations for 15 seconds and with an interval of 30 seconds.

In the participants of the intervention group, the calculation of the ideal tidal volume for each patient will be performed, after which they will be positioned in the supine position, the head elevated to 30º in assisted pressure-controlled ventilation mode, increasing 10 cmH2O in inspiratory pressure and, in assisted ventilation mode. controlled by volume, we will increase 50% of the tidal volume for a period of 10 minutes, observing the Ppeak that cannot exceed 40 cmH2O and the drive pressure that cannot exceed 15 cmH2O in both ventilation modes, and then a new aspiration will be performed. in the same way as the control group. The hemodynamics data will be taken from the multiparametric monitor of the hospitalization units (philips) and the respiratory mechanics data will be collected from the mechanical ventilator screen (Servo S; Drager; Newport), before and after the techniques. The volume of secretion will be stored in the collection flask (Water Seal 120 ml) and weighed using a high precision scale, discounting the weight of the collection flask.

The Informed Consent Form (ICF) will be signed by the responsible family member, containing information and explanations about the present study and the researcher will be available to explain doubts and questions at the time and afterwards through the telephone present at the ICF. All procedures will be performed under the supervision of the physiotherapist at the hospital. It is understood that this research may offer a minimal risk to volunteers, according to resolution 466/12 of the National Health Council, since they may have some discomfort and / or their hemodynamic situation altered by the application of the aforementioned physical therapy technique. As a counterpart, in case the predicted risk occurs, the subjects will receive all the necessary care from the researcher, together with the unit's physiotherapist and medical team, if necessary. The benefits to the subjects refer to the possibility of improving their respiratory function and bronchial hygiene.

ELIGIBILITY:
Inclusion Criteria:

* Interned in the Post-Operative Unit (UPO), Intensive Care Center (ICU) and Emergency.
* Using invasive mechanical ventilation for more than 48 hours.
* Hemodynamically stable (MAP 60-120 mmHg).

Exclusion Criteria:

* Diagnosis of ventilator-associated pneumonia.
* Individuals with pneumothorax and undrained hemothorax.
* Subcutaneous emphysema.
* Patients with peak pressure> 40 cmH2O.
* Patients diagnosed with neurological disease within 72 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
amount of secretion | 15 minutes after the technique.
  ml

SECONDARY OUTCOMES:
heart rate | Immediately before and after ande during the technique.
  bpm
respiratory rate | Immediately before and after and during the technique.
  bpm
mean arterial pressure systolic and dyastolic blood pressure | Immediately before and after ande during the technique.
  mmhg
peripheral saturation | Immediately before and after ande during the technique.
  SpO2 %
static compliance | Immediately before and after ande during the technique.
  ml/cmH2O
dynamic compliance | Immediately before and after ande during the technique.
  ml/cmH2O
current air volume | Immediately before and after ande during the technique.
  ml
peak pressure | Immediately before and after ande during the technique.
  cmH2O
plateau pressure | Immediately before and after ande during the technique.
  cmH2O
drive pressure | Immediately before and after ande during the technique.
  cmH2O

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Eibel, Dr, Principal Investigator — Instituto de Cardiologia
Locations (1):
- Instituto de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carvalho CR, Toufen C Jr, Franca SA. [Mechanical ventilation: principles, graphic analysis and ventilatory modalities]. J Bras Pneumol. 2007;33 Suppl 2S:S54-70. doi: 10.1590/s1806-37132007000800002. No abstract available. Portuguese. PMID 18026665
- [Result] Franca EE, Ferrari F, Fernandes P, Cavalcanti R, Duarte A, Martinez BP, Aquim EE, Damasceno MC. Physical therapy in critically ill adult patients: recommendations from the Brazilian Association of Intensive Care Medicine Department of Physical Therapy. Rev Bras Ter Intensiva. 2012 Mar;24(1):6-22. English, Portuguese. PMID 23917708
- [Result] Dennis DM, Jacob WJ, Samuel FD. A survey of the use of ventilator hyperinflation in Australian tertiary intensive care units. Crit Care Resusc. 2010 Dec;12(4):262-8. PMID 21143087
- [Result] Lemes DA, Zin WA, Guimaraes FS. Hyperinflation using pressure support ventilation improves secretion clearance and respiratory mechanics in ventilated patients with pulmonary infection: a randomised crossover trial. Aust J Physiother. 2009;55(4):249-54. doi: 10.1016/s0004-9514(09)70004-2. PMID 19929767
- [Result] Naue Wda S, Forgiarini Junior LA, Dias AS, Vieira SR. Chest compression with a higher level of pressure support ventilation: effects on secretion removal, hemodynamics, and respiratory mechanics in patients on mechanical ventilation. J Bras Pneumol. 2014 Jan-Feb;40(1):55-60. doi: 10.1590/S1806-37132014000100008. PMID 24626270
- [Result] Favretto DO, Silveira RC, Canini SR, Garbin LM, Martins FT, Dalri MC. Endotracheal suction in intubated critically ill adult patients undergoing mechanical ventilation: a systematic review. Rev Lat Am Enfermagem. 2012 Sep-Oct;20(5):997-1007. doi: 10.1590/s0104-11692012000500023. English, Portuguese, Spanish. PMID 23174846